CLINICAL TRIAL: NCT00966940
Title: The Efficacy and Safety of Travoprost, 0.004% Versus Tafluprost, 0.0015% in Primary Open-Angle Glaucoma or Ocular Hypertensive Patients
Brief Title: Efficacy and Safety of Travoprost 0.004% Versus Tafluprost 0.0015% in Patients With Primary Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SMA-08-16
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Glaucoma
Keywords: Glaucoma; IOP; Travoprost
MeSH Terms: conditions — Glaucoma | interventions — Travoprost; Ophthalmic Solutions; tafluprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost-to-tafluprost (Other): Travoprost first, with tafluprost second. Each product dosed for six weeks.
  Interventions: Drug: Travoprost 0.004% ophthalmic solution (TRAVATAN); Drug: Tafluprost 0.0015% ophthalmic solution
- Tafluprost-to-travoprost (Other): Tafluprost first, with travoprost second. Each product dosed for six weeks.
  Interventions: Drug: Travoprost 0.004% ophthalmic solution (TRAVATAN); Drug: Tafluprost 0.0015% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost 0.004% ophthalmic solution (TRAVATAN) — One drop in the qualifying eye(s) each evening at 6:00 PM for 6 weeks, topical administration
  Other Names: TRAVATAN
Drug: Tafluprost 0.0015% ophthalmic solution — One drop in the qualifying eye(s) each evening at 6:00 PM for 6 weeks, topical administration

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Travoprost 0.004% and Tafluprost 0.0015% in patients with primary open angle glaucoma or ocular hypertension when both medications are administered in the evening.

ELIGIBILITY:
Inclusion Criteria:

* An EC-reviewed and approved (for use in this study) informed consent form must be read, signed, and dated by the participating patient as well as signed and dated by the individual (Principal Investigator or other site personnel) obtaining the informed consent, before conducting the Screening Visit and prior to initiation of study procedures.
* Patients must be at least 21 years of age.
* Must be able to follow instructions and be willing and able to attend required study visits.
* Must have a clinical diagnosis of ocular hypertension or primary open-angle glaucoma in at least one eye (qualifying eye).
* Currently treated patients, in the investigator's judgment, should require a change in treatment for reasons of improved efficacy, tolerability or compliance.
* Must have IOP considered to be safe, in both eyes, in such a way that should assure clinical stability of vision and the optic nerve throughout the trial.
* Must have an intraocular pressure of > 21 mm Hg in at least one eye at 08:00 and > 19 mm Hg in the same eye at 16:00, and < 35 mm Hg in both eyes at all diurnal time points at Visit 2.
* Must have best corrected visual acuity of 6/60 (20/200 Snellen) or better in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Presence of other primary or secondary glaucomas not listed in inclusion criterion.
* Presence of extreme narrow angle with complete or partial closure in either eye, as measured by gonioscopy (occludable angles treated with a patent iridectomy are acceptable).
* Any abnormality preventing reliable applanation tonometry in qualifying eye(s).
* Any opacity or patient uncooperativeness that restricts adequate examination of the ocular fundus or anterior chamber of either eye.
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye. Blepharitis or non-clinically significant conjunctival injection is allowed.
* Intraocular conventional surgery or laser surgery in qualifying eye(s) less than three months prior to Visit 1.
* Risk of visual field or visual acuity worsening as a consequence of participation in the trial, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause apart from glaucoma.
* Women of childbearing potential not using reliable means of birth control, or pregnant or lactating females.
* Any clinically significant, serious, or severe medical or psychiatric condition.
* A condition, which in the opinion of the investigator, would interfere with optimal participation in the study, or which would present a special risk to the patient.
* Participation in any other investigational study within 30 days prior to Visit 2.
* Known medical history of allergy or sensitivity to any components of the preparations to be used in this trial that is deemed clinically significant in the opinion of the investigator.
* Use of systemic medications known to affect IOP (e.g., oral beta-adrenergic blockers,alpha-agonists and blockers, angiotensin converting enzyme inhibitors and calcium channel blockers), which have not been on a stable course for 7 days prior to Visit 2 or an anticipated change in the dosage during the course of the study.
* Anticipated use of systemic corticosteroids, by any route except inhaled, for greater than two weeks during the trial.
* A history of, or at risk for uveitis or cystoid macular edema (CME).
* History of ocular herpes simplex.
* Unwillingness to accept the risk of iris, skin, or eyelash changes associated with prostaglandin therapy.
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from four private practices located in Germany.
Groups:
- Travoprost-to-tafluprost: Travoprost, then tafluprost
- Tafluprost-to-travoprost: Tafluprost, then travoprost
Period: Period 1, First 6 Weeks
Arm/Group | Travoprost-to-tafluprost | Tafluprost-to-travoprost
Started | 28 | 23
Completed | 25 | 23
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 0
Period: Period 2, Second 6 Weeks
Arm/Group | Travoprost-to-tafluprost | Tafluprost-to-travoprost
Started | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost-to-tafluprost | Tafluprost-to-travoprost | Total
Number analyzed (Participants) | 28 | 23 | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 69.1 (7.8) | 68.5 (10.5) | 68.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP) at 8:00 PM
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 6 weeks
Population: This reporting group includes all patients randomized to both periods of the study and exposed to both study drugs.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Travoprost; Tafluprost: One drop in the qualifying eye(s) each evening at 6:00 PM for six weeks, administered topically
Arm/Group | Travoprost | Tafluprost
Number analyzed (Participants) | 48 | 48
mm Hg | 17.1 (3.17) | 17.7 (3.23)

2. Secondary Outcome: Mean Intraocular Pressure (IOP) at 8:00 AM
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 6 weeks
Population: This reporting group includes all patients randomized to both periods of the study and exposed to both study drugs.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Travoprost | Tafluprost
Number analyzed (Participants) | 48 | 48
mm Hg | 17.0 (2.36) | 17.5 (2.20)

3. Secondary Outcome: Mean Intraocular Pressure (IOP) at 10:00 AM
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 6 weeks
Population: This reporting group includes all patients randomized to both periods of the study and exposed to both study drugs.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Travoprost | Tafluprost
Number analyzed (Participants) | 48 | 48
mm Hg | 16.7 (2.39) | 17.3 (2.50)

4. Secondary Outcome: Mean Intraocular Pressure (IOP) at 12:00 PM
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 6 weeks
Population: This reporting group includes all patients randomized to both periods of the study and exposed to both study drugs.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Travoprost | Tafluprost
Number analyzed (Participants) | 48 | 48
mm Hg | 16.7 (2.47) | 17.2 (2.46)

5. Secondary Outcome: Mean Intraocular Pressure (IOP) at 2:00 PM
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 6 weeks
Population: This reporting group includes all patients randomized to both periods of the study and exposed to both study drugs.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Travoprost | Tafluprost
Number analyzed (Participants) | 48 | 48
mm Hg | 16.9 (2.69) | 17.3 (2.77)

6. Secondary Outcome: Mean Intraocular Pressure (IOP) at 4:00 PM
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 6 weeks
Population: This reporting group includes all patients randomized to both periods of the study and exposed to both study drugs.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Travoprost | Tafluprost
Number analyzed (Participants) | 48 | 48
mm Hg | 17.1 (2.85) | 17.6 (2.80)

7. Secondary Outcome: Mean Intraocular Pressure (IOP) at 6:00 PM
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 6 weeks
Population: This reporting group includes all patients randomized to both periods of the study and exposed to both study drugs.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Travoprost | Tafluprost
Number analyzed (Participants) | 48 | 48
mm Hg | 16.9 (3.12) | 17.6 (3.13)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 10-September-2009 to 2-March-2010.
Arm/Group | Travoprost | Tafluprost
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 0/51 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less